CLINICAL TRIAL: NCT07132515
Title: Efficacy and Safety of Anticoagulant Therapy for Portal Vein Thrombosis In Cirrhosis Patients With and Without Hepatocellular Carcinoma
Brief Title: Efficacy & Safety of Anticoagulants in Cirrhosis ± HCC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.23.07.2479
Record Dates: First submitted 2025-08-10; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis; HCC - Hepatocellular Carcinoma; Portal Vein Thrombosis
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular | interventions — Enoxaparin; apixaban

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anticoagulant in cirrhosis with HCC (Experimental): HCC patient on anticogulant like Enoxaparin (clexan), warfarrin(marivan), or DOAC(apixaban)
  Interventions: Drug: Enoxaparin, warfarrin, or apixaban
- Anticoagulant in Cirrhosis without HCC (Experimental): Benign thrombus in cirrhotic patient on anticoagulant like Enoxaparin (clexan), warfarrin(marivan), or DOAC(apixaban)
  Interventions: Drug: Enoxaparin, warfarrin, or apixaban
- No anticoagualnt in Cirrhosis with or without HCC (No Intervention): cirrhotic patients with thrombosis with or without HCC not on anticoagulant

INTERVENTIONS:
Drug: Enoxaparin, warfarrin, or apixaban — Enoxaparin, warfarrin, or apixaban
  Arms: Anticoagulant in Cirrhosis without HCC; Anticoagulant in cirrhosis with HCC

SUMMARY:
We will give an anticoagulant against portal vein thrombosis, and watch for the results.

ELIGIBILITY:
Inclusion Criteria:

* Portal vein thrombosis, Cirrhosis, With or without HCC, Child A & B

Exclusion Criteria:

* Platelets<10000, Createnine >1.9, Budd ciarri, Uncontrolled active bleeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Portal vein thrombosis | 6 months
  determine if thrombus resolved or not on anticcoagulant by triphasic CT

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
when this clinical trial will be finished and have the results